CLINICAL TRIAL: NCT01940419
Title: Peroperative Tranexamic Acid as Prophylaxis of Haemorrhage in Benign Hysterectomy - a Randomized, Placebo-controlled Trial
Brief Title: Testing of the Drug Tranexamic Acids as Prophylaxis of Bleeding in Benign Surgical Removal of the Uterus
Acronym: PeTraH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hillerod Hospital, Denmark (Other)
Collaborators: Rigshospitalet, Denmark (Other); Odense University Hospital (Other); Central Denmark Region (Other); Research grant from Nordsjællands Hospital (Unknown); The fund of Olga Bryde (Unknown); The Danish hysterectomy and hysteroscopy database (Unknown)
Responsible Party: Principal Investigator, Märta Fink Topsøe, DM, PhD-student, Hillerod Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2011-425; 2012-005407-40 (EudraCT Number)
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Gynecologic Surgical Procedures; Hysterectomy; Tranexamic Acid
Keywords: Reduction of blood loss; Surgical complication; Hysterectomy; Antifibrinolytic Agents; Randomized Controlled Trials
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (Active Comparator): 1g Tranexamic acid iv just before surgery
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): sterile sodium chloride 9mg/ml iv
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — 1g Tranexamic acid iv administered over 10 minutes just before surgery
  Other Names: Cyklokapron
  Arms: Tranexamic Acid
Drug: Placebo — 10 ml sodium chloride iv administered over 10 minutes just before surgery
  Arms: Placebo

SUMMARY:
In Denmark, 4400 women annually undergo hysterectomy on benign background (surgical removal of the uterus). 10% of these women experience bleeding complications. The drug Tranexamic Acid (Cyklokapron) has showed significant reduction of bleeding in relation to other types of surgery. The hypothesis of this study is that Tranexamic Acid could also reduce the operative bleeding associated with benign hysterectomy. The study will be carried out as a randomized, placebo-controlled national multicenter trial

DETAILED DESCRIPTION:
In Denmark, there are approximately 4400 elective benign hysterectomies annually. In about 10% of these there will occur a per- or postoperative bleeding complications with increased hospital stay, reoperations and prolonged sick leave as a result. The pharmaceutical product 'Tranexamic acid' has proved to be effective in reducing blood loss in other forms of surgery, in trauma patients, and in relation to certain medical conditions. The hypothesis of the proposed study is that Tranexamic acid could also reduce the operative bleeding associated with hysterectomy on benign indications. Based on the literature and previous studies, the objective of the trial is an average bleeding reduction of 25%.

The clinical trial will be conducted as a randomized, placebo-controlled, double blind multicenter trial in gynecological departments several places in Denmark: Nordsjællands Hospital, Rigshospitalet, Odense University Hospital and Aarhus University Hospital - Skejby. The subjects will be recruited in outpatient clinics of the gynecological departments. During the study there will be an ongoing monitoring by external partner. The experiment is approved by all relevant bodies. The total period of time in which the trial is planned to last is one year commencing 01.02.3013 and ending 28.02.2014. All together the trial will include 314 participants determined by presumed bleeding reduction, the average bleeding on hysterectomy and type 1 error of 0.05 and type 2 error of 0.20. Randomization will be conducted electronically and both clinician, patient and data collector we will be blinded. Data for the study will partly be collected through registrations to the already well established and well functioning Danish Hysterectomy and Hysteroscopy Database. Data used in relation to the study will be validated by examining the manual records in conjunction with data extraction. The results will be analyzed by univariate and multivariate analyzes and static regression analyzes. All final results from the study will be sought published in recognized international journals.

Regarding ethical aspects it is noted that the study is carried out with the highest standard of design, and with a proven drug without unexpected side effects or disadvantages. In the literature, there seems no evidence to suspect an increased risk of blood clot formation using the drug. However, it seems clear that the incidence of complications associated with hysterectomy is quite high. It is therefore ethically fully responsible and appropriate to carry out the planned study with the desire to ensure the quality and improve hysterectomy, surgery.

The project is supported by funds and receives no commercial support.

ELIGIBILITY:
Inclusion Criteria:

• Women over 18 who is to undergo elective benign hysterectomy

Exclusion Criteria:

* Known thrombophilia
* Active / previous thromboembolic disease
* Family history of thromboembolic disease (thrombophilia in the family)
* Hypersensitivity to any ingredient in Tranexamic acid
* Renal impairment
* Ongoing hematuria
* Subarachnoid hemorrhage
* Daily use of any type of blood thinners (Clopidogrel / Marevan / Warfarin / Nonsteroidal Antiinflammatory Drugs (not when pain is the indication))
* Preoperative use of Tranexamic acid within 24 hours of the operation
* Known malignancy or hysterectomy as part of the investigation for suspected malignancy
* Insufficient understanding of the information concerning the project: language disabilities, intellectual limitations, or the like.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Intraoperative bleeding | 1 day (Bleeding is measured immediately after surgery)
  In relation to the trial there is at set of standards to objectify blood loss during surgery. Output and input will be weighed and will form the basis of the calculated operative blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Märta F Topsøe, DM, Principal Investigator — Department of gynecology and obstetrics, Nordsjællands Hospital, 3400 Hillerød
Locations (1):
- Department of gynecology and obstetrics, Nordsjællands Hospital, Hillerød, Denmark

REFERENCES:
- [Background] Henry DA, Carless PA, Moxey AJ, O'Connell D, Stokes BJ, Fergusson DA, Ker K. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2011 Mar 16;2011(3):CD001886. doi: 10.1002/14651858.CD001886.pub4. PMID 21412876
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Lethaby A, Farquhar C, Cooke I. Antifibrinolytics for heavy menstrual bleeding. Cochrane Database Syst Rev. 2000;(4):CD000249. doi: 10.1002/14651858.CD000249. PMID 11034679
- [Background] Dunn CJ, Goa KL. Tranexamic acid: a review of its use in surgery and other indications. Drugs. 1999 Jun;57(6):1005-32. doi: 10.2165/00003495-199957060-00017. PMID 10400410
- [Background] Sukeik M, Alshryda S, Haddad FS, Mason JM. Systematic review and meta-analysis of the use of tranexamic acid in total hip replacement. J Bone Joint Surg Br. 2011 Jan;93(1):39-46. doi: 10.1302/0301-620X.93B1.24984. PMID 21196541
- [Background] Astedt B, Liedholm P, Wingerup L. The effect of tranexamic acid on the fibrinolytic activity of vein walls. Ann Chir Gynaecol. 1978;67(6):203-5. PMID 742821
- [Background] Lukes AS, Moore KA, Muse KN, Gersten JK, Hecht BR, Edlund M, Richter HE, Eder SE, Attia GR, Patrick DL, Rubin A, Shangold GA. Tranexamic acid treatment for heavy menstrual bleeding: a randomized controlled trial. Obstet Gynecol. 2010 Oct;116(4):865-875. doi: 10.1097/AOG.0b013e3181f20177. PMID 20859150
- [Background] Bonnar J, Sheppard BL. Treatment of menorrhagia during menstruation: randomised controlled trial of ethamsylate, mefenamic acid, and tranexamic acid. BMJ. 1996 Sep 7;313(7057):579-82. doi: 10.1136/bmj.313.7057.579. PMID 8806245
- [Background] Coulter A, Kelland J, Peto V, Rees MC. Treating menorrhagia in primary care. An overview of drug trials and a survey of prescribing practice. Int J Technol Assess Health Care. 1995 Summer;11(3):456-71. doi: 10.1017/s0266462300008679. PMID 7591547